CLINICAL TRIAL: NCT07314060
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial Evaluating the Efficacy and Safety of TQH2929 Injection in Patients With Acute Exacerbations of Generalized Pustular Psoriasis
Brief Title: A Clinical Trial of TQH2929 Injection in Patients With Acute Flare-up of Generalized Pustular Psoriasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQH2929-II-01
Record Dates: First submitted 2025-12-15; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-10

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQH2929 Injections (Experimental): Intravenous infusion, single dose
  Interventions: Drug: TQH2929 Injections
- TQH2929 Placebo (Placebo Comparator): Intravenous infusion, single dose
  Interventions: Drug: TQH2929 Placebo

INTERVENTIONS:
Drug: TQH2929 Injections — TQH2929 is a humanized monoclonal antibody that interfering with the signal cascade.
  Arms: TQH2929 Injections
Drug: TQH2929 Placebo — Placebo contains no active substance.
  Arms: TQH2929 Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase II clinical study, all subjects need to use TQH2929 injection/placebo. The aim was to demonstrate the efficacy and safety of TQH2929 injection in patients with acute exacerbations of generalized pustular psoriasis, with a total of 36 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 or ≤75 years old at screening, regardless of gender;
* Meet the diagnostic criteria defined by the 2017 European Society for Clinical Nutrition and Metabolism (ESPEN) Research Workshop (ERASPEN) consensus and be diagnosed as （generalized pustular psoriasis(GPP);
* Compliant with GPP acute onset;
* Able to read and understand, and willing to sign the informed consent form;
* Willing and compliant with study visits and related procedures;
* Female subjects of childbearing age should agree that contraceptive measures must be used during the study and for 6 months after the end of the study;

Exclusion Criteria:

* Pustules are limited to psoriasis vulgaris on psoriasis plaques;
* Concomitant skin disease or medical disease that may interfere with the investigator's evaluation of the subject's treatment response;
* Presence of severe, progressive, or uncontrolled disease, or signs and symptoms that are not suitable for participation in the investigator, in the judgment of the investigator:
* Serum virological abnormalities during the screening period;
* Chest radiology examination shows that the subject has active tuberculosis or a history of contact with open tuberculosis subjects in the past 6 months or a positive Interferon-Gamma Release Assays(IGRA) test;
* History of serious infection leading to hospitalization within 2 months prior to baseline;
* Active infection requiring systemic antibiotics, systemic antifungals, or systemic antiviral therapy within 2 weeks prior to baseline, according to the investigator's assessment;
* History of opportunistic infection within 6 months prior to baseline;
* Received live (attenuated) vaccine treatment within 12 weeks prior to baseline;
* Any major surgery within 4 weeks prior to baseline or planned major surgery during the study;
* Received blood transfusion within 4 weeks prior to baseline;
* Participated in clinical trials of other drugs or medical devices within 4 weeks before baseline;
* Any known or suspected congenital or acquired immunodeficiency state or condition that may compromise the subject's immune status;
* Subjects with any type of active malignancy or a history of malignancy;
* Alcohol, drug and known drug dependence;
* Pregnant or lactating women;
* Subjects cannot tolerate intravenous infusion administration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a score of 0 for the pustule subterm | 1 week
  Percentage of patients with a Physician's Global Assessment of Generalized Pustular Psoriasis (GPPGA) pustular subitem of 0 (no visible pustules) at week 1 among all enrolled patients.

SECONDARY OUTCOMES:
Percentage of patients with a Generalized Pustular Psoriasis Physician Global Assessment(GPPGA) total score of 0 or 1 | 1 week and 4 weeks
  Percentage of patients with a total Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) score of 0 (clear) or 1 (almost clear) at weeks 1 and 4.
Percentage change from baseline in Generalized Pustular Psoriasis Area and Severity Index (GPPASI) total score | 1 week and 4 weeks
  Percentage change from baseline in the total score of generalized pustular psoriasis area and severity index (GPPASI) at week 1 and week 4.
Change from baseline in Generalized Pustular Psoriasis Area and Severity Index(GPPASI) total score | 1 week and 4 weeks
  Change from baseline in Generalized Pustular Psoriasis Area and Severity Index(GPPAS) total score at week 1 and week 4. If lower than the baseline score, indicate a certain degree of disease relief; conversely, if higher, it indicates an aggravation of the disease symptoms.
Percentage of patients with Generalized Pustular Psoriasis Area and Severity Index(GPPASI) 50 | 1 week and 4 weeks
  Percentage of patients who achieved Generalized Pustular Psoriasis Area and Severity Index(GPPASI) 50 at week 1 and week 4.
Percentage of patients with Generalized Pustular Psoriasis Area and Severity Index(GPPASI) 75 | 1 week and 4 weeks
  Percentage of patients who achieved Generalized Pustular Psoriasis Area and Severity Index(GPPASI) 75 at week 1 and week 4
Percentage of patients with pustule subterm achieving a score of 0 | 4 weeks
  Percentage of patients with Generalized Pustular Psoriasis Physician Global Assessment(GPPGA) pustule subterm achieving a score of 0 (no visible pustules) at week 4.
Change from baseline in Psoriasis Symptom Scale (PSS) score | 4 weeks
  Change from baseline in Psoriasis Symptom Scale (PSS) score at week 4
Change from baseline in disease life quality index (DLQI) | 4 weeks
  Change from baseline in skin disease life quality index (DLQI) at week 4. If lower than the baseline score, indicate a certain degree of disease relief; conversely, if higher, it indicates an aggravation of the disease symptoms.
Adverse Drug Event (AE) | 113 days or 169 days
  Any untoward medical occurrence of a subject following drug treatment or exposure to an experimental factor, whether or not causally related to treatment or exposure.
Serious Adverse Event (SAE) | 113 days or 169 days
  An event that occurs in the course of a clinical trial that results in the death of a subject or patient, serious deterioration in health, hospitalization or prolongation of hospitalization, permanent disability or loss of function, or serious consequences such as birth defects or birth defects.
Treatment-Emergent Adverse Events (TEAES) | 113 days or 169 days
  Adverse events that occur during treatment, including from the start of treatment to a certain period of time after the end of treatment, may be directly or indirectly related to treatment.
Abnormal clinical laboratory examination indicators | 113 days or 169 days
  Any laboratory abnormalities that occur during the test.
Time of maximum concentration (Tmax) | 1 hour pre-dose on day 1, immediately post dose, 1, 6, 24, 48, 168, 336, 504, 672, 1344, 2016, 2688 hours post dose. Day 8 Immediately after the end of salvage therapy administration, 1, 6, 24, 48 hours post dose
  It refers to the time it takes for the human blood concentration curve to reach the highest concentration (peak concentration) after a single dose, measured in hours or minutes.
Maximum Concentration (Cmax) | 1 hour pre-dose on day 1, immediately post dose, 1, 6, 24, 48, 168, 336, 504, 672, 1344, 2016, 2688 hours post dose. Day 8 Immediately after the end of salvage therapy administration, 1, 6, 24, 48 hours post dose
  The highest blood concentration reached after the drug is absorbed in the body.
Area Under the Curve (AUC) | 1 hour pre-dose on day 1, immediately post dose, 1, 6, 24, 48, 168, 336, 504, 672, 1344, 2016, 2688 hours post dose. Day 8 Immediately after the end of salvage therapy administration, 1, 6, 24, 48 hours post dose
  It refers to the area covered by the concentration of a drug in the blood under the curve of changes over time.
Apparent Volume of Distribution(Vd/F) | 1 hour pre-dose on day 1, immediately post dose, 1, 6, 24, 48, 168, 336, 504, 672, 1344, 2016, 2688 hours post dose. Day 8 Immediately after the end of salvage therapy administration, 1, 6, 24, 48 hours post dose
  When the drug reaches dynamic equilibrium in the body, the ratio of the amount of drug in the body to the blood concentration is called the apparent volume of distribution.
Apparent Clearance (CL/F) | 1 hour pre-dose on day 1, immediately post dose, 1, 6, 24, 48, 168, 336, 504, 672, 1344, 2016, 2688 hours post dose. Day 8 Immediately after the end of salvage therapy administration, 1, 6, 24, 48 hours post dose
  The sum of drug clearance rates of liver and kidney, etc.
Plasma half-life time (t1/2) | 1 hour pre-dose on day 1, immediately post dose, 1, 6, 24, 48, 168, 336, 504, 672, 1344, 2016, 2688 hours post dose. Day 8 Immediately after the end of salvage therapy administration, 1, 6, 24, 48 hours post dose
  The time it takes for the concentration of the drug in the plasma to drop by half.
Anti-drug antibody (ADA) | Through study completion, an average of half a year
  Incidence of anti-drug antibodies (ADA) in subjects.

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - Peking University First Hospita, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Southern Medical University Dermatology Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Henan University of science and technology, Luoyang, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The fifth Affiliated hospital of zhengzhou university, Zhengzhou, Henan
  - Shiyan Renmin Hospital, Shiyan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The General Hospital Of Hunan University Of Medicine, Huaihua, Hunan
  - The first hospital of jilin university, Changchun, Jilin
  - The first hospital of china medical university, Shenyang, Liaoning
  - Shandong First Medical University Affiliated Dermatology Hospital, Jinan, Shandong
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People' s Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Jiaxing First Hospital, Jiaxing, Zhejiang
  - The first affiliated hospital of ningbo university, Ningbo, Zhejiang